CLINICAL TRIAL: NCT07289048
Title: A Prospective, Single-Arm, Exploratory Clinical Study of IBI363 in Patients With Extensive-Stage Small Cell Lung Cancer (ES-SCLC) Following Progression on Immunotherapy
Brief Title: A Prospective, Single-Arm, Exploratory Study of IBI363 in ES-SCLC Patients After Immunotherapy Progression
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Xiaorong Dong, Professor, Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ES-SCLC-IIT-01
Record Dates: First submitted 2025-12-05; First posted 2025-12-17 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: SCLC,Extensive Stage

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- IBI363（PD-1/IL-2a-bias） (Experimental)
  Interventions: Drug: IBI363（PD-1/IL-2a-bias）

INTERVENTIONS:
Drug: IBI363（PD-1/IL-2a-bias） — The administration route of IBI363 is intravenous infusion. Based on the cumulative safety data of IBI363 monotherapy, the administration protocol of IBI363 adopts the Priming design. The subjects will receive 1 dose of 100 μg/kg (initial dose) of IBI363 on the first day of the first cycle (C1D1), aIBI363（PD-1/IL-2a-bias）nd then the target dose of 3 mg/kg Q3W IBI363 will be administered starting 7 days later. The administration period except for the first cycle is 21 days (the first cycle lasts for 28 days).

SUMMARY:
This study is a prospective, single-arm, exploratory clinical trial designed to evaluate the efficacy and safety of IBI363 in patients with extensive-stage small cell lung cancer (ES-SCLC) who have progressed after at least two prior lines of standard therapy, including PD-1/PD-L1 inhibitor-based immunotherapy. A total of 35 patients were enrolled. The primary endpoint is the objective response rate (ORR), as assessed by investigators according to RECIST 1.1 criteria. Following a screening period of up to 28 days, patients will receive IBI363 treatment until disease progression, onset of intolerable toxicity, withdrawal of informed consent, completion of 24 months of therapy, discontinuation due to other protocol-specified reasons, or early termination of the study.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 to 75 years (inclusive), male or female.
2. Histologically confirmed small cell lung cancer (SCLC).
3. Extensive-stage SCLC refractory to 2 to 3 prior lines of systemic anti-tumor therapy, which must have included PD-1/PD-L1 immunotherapy.
4. At least one measurable target lesion as per RECIST 1.1 criteria. The target lesion must be measurable (longest diameter ≥10 mm at baseline, or for lymph nodes, short-axis diameter ≥15 mm) and not have been previously irradiated, or have demonstrated clear progression after local therapy. Lesions solely within the brain are not acceptable as target lesions.
5. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
6. Life expectancy ≥ 3 months.
7. Adequate organ function,
8. Fertile patients (male and female) must agree to use highly effective contraception (e.g., hormonal, barrier methods, or abstinence) with their partner during the trial and for at least 6 months after the last dose. A serum pregnancy test for women of childbearing potential must be negative within 7 days prior to the first study dose.
9. Subjects must provide written informed consent before initiating any study-specific procedures.

Exclusion Criteria:

1. Histological diagnosis of combined small cell lung cancer (e.g., mixed SCLC and NSCLC), transformed non-small cell lung cancer (e.g., SCLC transformed from NSCLC), or transformed SCLC (e.g., NSCLC transformed to SCLC).
2. Known history of hypersensitivity (≥ Grade 3 per CTCAE v5.0) to any antibody-based therapeutic agent, or known hypersensitivity to the active substance or inactive excipients of the investigational product.
3. Major surgical procedure (excluding needle biopsy) or significant trauma within 4 weeks prior to the first dose of study treatment, or anticipation of the need for elective surgery during the study period.
4. Systemic corticosteroid therapy (>10 mg/day prednisone or equivalent) within 14 days prior to the first dose of study treatment, with the following exceptions: topical, ocular, intra-articular, intranasal, or inhaled corticosteroids; short-term prophylactic use (e.g., for contrast media allergy); or treatment with other immunosuppressive agents within 4 weeks.
5. Use of immunomodulatory drugs (e.g., thymosin, interleukin-2, interferon) within 14 days prior to the first dose of study treatment.
6. Administration of a live attenuated vaccine within 4 weeks prior to the first dose of study treatment.
7. Prior allogeneic hematopoietic stem cell transplantation or solid organ transplantation.
8. Adverse events from prior anti-tumor therapy have not recovered to ≤ Grade 1 per CTCAE v5.0 or the levels specified in the inclusion criteria (with the exception of toxicities deemed not to pose a safety risk by the investigator, such as alopecia, Grade 2 peripheral neuropathy, or hypothyroidism stable on hormone replacement therapy).
9. Untreated brain metastases (subjects with treated brain metastases are eligible if clinically stable for ≥4 weeks prior to the first dose, off steroid therapy for ≥2 weeks, and without significant peritumoral edema on imaging); leptomeningeal metastasis or brainstem metastasis; spinal cord compression (radiologically identified, regardless of symptoms).
10. Active infection requiring intravenous anti-infective therapy at the time of screening.
11. History of immunodeficiency, including a positive test for human immunodeficiency virus (HIV).
12. Active hepatitis B (HBsAg positive and HBV-DNA ≥1000 IU/mL or copies/mL) or active hepatitis C (HCV antibody positive and HCV RNA above the upper limit of normal).
13. Interstitial lung disease (except for radiation-induced fibrosis not requiring corticosteroid therapy).
14. Significant cardiovascular and cerebrovascular disease history
15. Active autoimmune disease, or history of autoimmune disease with potential for recurrence (exceptions include well-controlled autoimmune thyroiditis, type I diabetes, vitiligo, childhood atopic dermatitis resolved, psoriasis not requiring systemic therapy in the past 2 years, etc.).
16. Prior history of ≥ Grade 3 immune-related adverse event (irAE) or ≥ Grade 2 immune-related myocarditis associated with prior immunotherapy.
17. History of other malignancies, except for those cured for ≥2 years, such as non-melanoma skin cancer, localized prostate cancer, or carcinoma in situ (e.g., cervical carcinoma in situ).
18. Pleural effusion or ascites requiring therapeutic intervention (subjects with stable effusion not requiring drainage or stable for ≥1 week after drainage may be eligible); pericardial effusion (asymptomatic, minimal effusion not requiring intervention per investigator's assessment is allowed). If intra-cavitary anti-tumor agents were used during drainage, a washout period of at least 5 half-lives or 21 days (whichever is shorter) must be completed prior to the first dose.
19. Known history of alcohol or drug dependence.
20. History of psychiatric disorders or anticipated poor compliance.
21. Pregnancy or lactation.
22. Any other condition deemed by the investigator to potentially compromise the subject's safety or compliance, or make the subject unsuitable for the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2025-12-20 (Estimated); Primary Completion 2027-12-30 (Estimated); Study Completion 2028-12-30 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | every 12 weeks (±7 days) up to 2 years
  Objective response rate (ORR) is deﬁned as the rate of patients, among all those enrolled,who achieve a best overall response [complete response (CR) or partial response (PR)] according to the RECIST v1.1 across all post-enrolment time-points until the end of follow up for disease progression.

SECONDARY OUTCOMES:
Progression-free survival (PFS) | Up to approximately 24 months.
  Progression-free survival (PFS) is deﬁned as the time from the date of enrolment until documented progression (according to RECIST v1.1) or death if progression is not documented.
overall survival（OS） | Up to approximately 24 months.
  Overall Survival (OS) is defined as the time from first dose of study treatment) until death from any cause.
AE | Up to approximately 24 months.
  Adverse events (AEs) according to CTCAE v5.0 (any-cause as well as treatment-related) including AEs leading to dose delays and/or interruptions, withdrawal of protocol treatment, and death.

IPD SHARING:
Plan to Share IPD: No